CLINICAL TRIAL: NCT04139148
Title: Study on the Effectiveness of "Treatment Regulation Mode" Based on Neuromodulation and Electronic Follow-up to Reduce Relapse Behavior in Patients With Substance Dependence
Brief Title: Transcranial Direct Current Stimulation (tDCS) Combined With Computerized Cognitive Addiction Therapy(CCAT) and, Electronic Follow-up for Methamphetamine(MA) Dependent Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Mental Health Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NZhong-002
Record Dates: First submitted 2019-04-12; First posted 2019-10-25 (Actual); Last update posted 2019-11-18 (Actual); Status verified 2019-10

CONDITIONS: Methamphetamine-dependence; Transcranial Direct Current Stimulation; Computerized Cognitive AddictionTherapy; Electronic Health Records

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- True tDCS Combined With CCAT (Active Comparator): Ture transcranial direct current stimulation (tDCS) intervention combined with computerized cognitive addiction therapy(CCAT) group, last 25 minutes per day for 4 weeks(5 days/week). Electronic follow-up for 6 month including drug knowledge every week, self-evaluation every two weeks and outpatient follow-up reminder every four weeks.
  Interventions: Device: Ture Transcranial Direct Current Stimulation (tDCS)
- Sham tDCS Combined With CCAT (Sham Comparator): Sham transcranial direct current stimulation (tDCS) intervention combined with computerized cognitive addiction therapy(CCAT) group, last 25 minutes per day for 4 weeks(5 days/week). Electronic follow-up for 6 month including only outpatient follow-up reminder every four weeks.
  Interventions: Device: Sham Transcranial Direct Current Stimulation (tDCS)
- Control group (No Intervention): During the treatment, the participants in control group only received treatment such as education of psychology, health and judicature, physical training as well as vocational training as usual in the compulsory rehabilitation center.

INTERVENTIONS:
Device: Ture Transcranial Direct Current Stimulation (tDCS) — Ture 1-2 mA current of tDCS intervention in patients' binary brain DLPFC areas(20 mm).
  Arms: True tDCS Combined With CCAT
Device: Sham Transcranial Direct Current Stimulation (tDCS) — Sham tDCS intervention in patients' binary brain DLPFC areas(20 mm).
  Arms: Sham tDCS Combined With CCAT

SUMMARY:
Transcranial direct current stimulation (tDCS) combined with computerized cognitive addiction therapy(CCAT) for methamphetamine(MA) dependent patients in voluntary drug rehabilitation center. Electronic medical systems were applied for drug related knowledge education, self-evaluation and outpatient follow-up reminder after intervention in order to reduce relapse behaviors.

ELIGIBILITY:
Inclusion Criteria:

* Methamphetamine dependent patients with normal eyesight and hearing.

Exclusion Criteria:

* any diagnosis of DSM-IV axis I diseases.
* any physical diseases which might influence cognitive function such as epilepsy, cerebrovascular disease or brain injury.
* negative behaviors or harm to others.
* cognitive enhance drug use history in last 6 months.
* other drug dependence(except nicotine).

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2019-02-01 (Actual); Primary Completion 2020-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline cue-induced craving at 2 weeks | 2 weeks
  Participants were instructed to watch methamphetamine-related videos by VR and rate their level of craving after smelling and recalling the last time they engaged in drug use. Craving was assessed by visual analog scales (VAS), with 0 mm being "no craving"and 100 mm representing "most craving ever experienced for methamphetamine".
Change from Baseline cue-induced craving at 4 weeks | 4 weeks
  Participants were instructed to watch methamphetamine-related videos by VR and rate their level of craving after smelling and recalling the last time they engaged in drug use. Craving was assessed by visual analog scales (VAS), with 0 mm being "no craving"and 100 mm representing "most craving ever experienced for methamphetamine".

SECONDARY OUTCOMES:
Attention bias towards methamphetamine | 2 weeks，4 weeks
  A Chinese version of the MA addiction dot probe task (DPT) is used to evaluate the attention bias towards drugs.
cognitive function | 2 weeks，4 weeks
  Chinese version of the CogState Battery was used to assess cognitive function.
response inhibition function | 2 weeks，4 weeks
  stop signal task
reward-related function | 2 weeks，4 weeks
  Delay Discounting Task

CONTACTS AND LOCATIONS:
Overall Officials: Na Zhong, doctor, Principal Investigator — Shanghai Mental Health Center
Locations (1):
- Shanghai Mental Health Center, Shanghai, China

IPD SHARING:
Plan to Share IPD: Undecided